CLINICAL TRIAL: NCT02006524
Title: Screening for Silent Atrial Fibrillation During Influenza Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Monika Hollander, MD, PhD, MD PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-85
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Atrial Fibrillation
Keywords: Silent atrial fibrillation; primary care; screening; influenza vaccination
MeSH Terms: conditions — Atrial Fibrillation; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Screening with MyDiagnostick (Active Comparator): All patients eligible for influenza vaccination are screened for atrial fibrillation with the MyDiagnostick, an easy to use and patient friendly device.
  Interventions: Device: 'MyDiagnostick

INTERVENTIONS:
Device: 'MyDiagnostick

SUMMARY:
Silent atrial fibrillation is an important cause of unnecessary strokes. If diagnosed and treated in time with anticoagulants, many disabling strokes can be prevented. In order to improve the diagnosis of atrial fibrillation the MyDiagnostick is developed; a user friendly and easy to use stick that diagnoses atrial fibrillation in one minute. During influenza vaccination, many patients who are also at risk for atrial fibrillation visit the general practice. This offers an ideal opportunity for screening for atrial fibrillation. The study investigates the yield of screening for atrial fibrillation with the MyDiagnostick during influenza vaccination (newly detected atrial fibrillation with corresponding CHA2DS2-Vasc score).

ELIGIBILITY:
Inclusion Criteria:

* Eligible for influenza vaccination

Exclusion Criteria:

* Not eligible for influenza vaccination

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3269 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Newly detected AF | during influenza vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Robert Tieleman, MD PhD, Principal Investigator — Martini Ziekenhuis Groningen; Monika Hollander, MD PhD, Principal Investigator — Julius Center UMC Utrecht
Locations (1):
- General Practices, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] Kaasenbrood F, Hollander M, Rutten FH, Gerhards LJ, Hoes AW, Tieleman RG. Yield of screening for atrial fibrillation in primary care with a hand-held, single-lead electrocardiogram device during influenza vaccination. Europace. 2016 Oct;18(10):1514-1520. doi: 10.1093/europace/euv426. Epub 2016 Feb 6. PMID 26851813